CLINICAL TRIAL: NCT03515499
Title: Incentives for Medication Adherence in Adolescents With Asthma
Brief Title: Incentives for Adherence in Adolescent Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-0089
Record Dates: First submitted 2018-02-05; First posted 2018-05-03 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Asthma; Asthma in Children
Keywords: Adherence; Incentives
MeSH Terms: conditions — Asthma | interventions — Fertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Active Comparator): The control arm will have medication monitoring sensors placed on their asthma medications. They will have reminders to take their medicines and access to a mobile app that will show them trends in their medication use.
  Interventions: Behavioral: Medication device monitoring and reminders
- Treatment arm (Experimental): The treatment arm will have medication monitoring sensors placed on their asthma medications. They will have reminders to take their medicines and access to a mobile app that will show them trends in their medication use. Additionally, they will be paid up to $1 per day for perfect medication adherence.
  Interventions: Behavioral: Incentives; Behavioral: Medication device monitoring and reminders

INTERVENTIONS:
Behavioral: Incentives — Subjects in the treatment arm will be paid up to $1 per day over 3 months for perfect medication adherence. Adherence rates will then be compared between the 2 groups.
  Arms: Treatment arm
Behavioral: Medication device monitoring and reminders — Bluetooth enabled sensor device for medication reminders, as well as mobile app to track medication use.

SUMMARY:
Financial incentives have been suggested as a possible means for increasing adherence to asthma medications. This study will evaluate an incentive strategy (daily small reward for adherence) in maintaining high levels of adherence as tracked by adherence sensors in adolescents with asthma.

DETAILED DESCRIPTION:
Two groups will be enrolled. The control group will have mediation monitoring sensors placed on their controller inhalers. The treatment group will also have the monitoring sensors placed on their medications, however they will be paid up to $1 per day for perfect adherence for 3 months. Both groups will be monitored for 4 months. 10 subjects will be chosen from each group to complete semi-structured phone interviews

ELIGIBILITY:
Inclusion Criteria:

* physician diagnosed asthma
* on at least one inhaled controller medication

Exclusion Criteria:

* language other than English or Spanish (these are the only languages supported by the adherence monitoring application)
* other severe chronic lung disease including tracheostomy/ventilator dependence, interstitial lung disease or cystic fibrosis, or significant developmental delay.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2018-07-06 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
Change in adherence rates | Daily for 12 weeks
  This Outcome will measure the difference in adherence at the end of the study period between the 2 groups as measured by the adherence devices (calculated as percent adherence per week over the 12 week study period).

SECONDARY OUTCOMES:
Changes in Qualitative outcomes - Barriers | After 3 months of monitoring
  Qualitative methodology will be used to evaluate patient attitudes towards the incentive program, as well as barriers of adherence, using semi-structured interviews. The investigators will obtain information on attitudes regarding barriers to medication adherence
Changes in Qualitative outcomes - Facilitators | After 3 months of monitoring
  Qualitative methodology will be used to evaluate patient attitudes towards the incentive program, as well as facilitators of adherence, using semi-structured interviews. The investigators will obtain information on attitudes regarding facilitators to adequate medication adherence.
Changes in Qualitative outcomes - Incentives | After 3 months of monitoring
  Qualitatively assessed feelings regarding incentives
  Qualitative methodology will be used to evaluate patient feelings towards the incentive program.The investigators will obtain information on incentives to adequate medication adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Hoch, MD, Principal Investigator — Assistant Professor
Locations (1):
- Childrens Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers

REFERENCES:
- [Derived] Keyser HH, Brinton JT, Bothwell S, Camacho M, Kempe A, Szefler SJ. Encouraging adherence in adolescents with asthma using financial incentives: An RCT. Pediatr Pulmonol. 2023 Oct;58(10):2823-2831. doi: 10.1002/ppul.26594. Epub 2023 Jul 14. PMID 37449768